CLINICAL TRIAL: NCT07308080
Title: Combined Effects of Near-Infrared Light and Vibration on Pain, Sleep Quality and Symptoms Severity in Diabetic Patients With Restless Leg Syndrome
Brief Title: Combined Effects of Near-Infrared Light and Vibration on Diabetic Patients With Restless Leg Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/038
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Restless Leg Syndrome (RLS)
Keywords: RLS, Diabetic patient, Near-Infrared Light, Vibration, Pain, Sleep Quality
MeSH Terms: conditions — Restless Legs Syndrome; Pain; Sleep Initiation and Maintenance Disorders | interventions — Vibration

STUDY DESIGN:
Intervention Model Description: After recruitment of participants into the study, they will be allocated to their respective group utilizing the online randomization tool.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A( Vibration Therapy + Conventional Physical Therapy) (Experimental): Participants allocated to this group will receive vibration therapy in addition to conventional physical therapy. Localized vibration will be applied to the calf muscles using a low-voltage vibration device for 10 minutes during supervised rehabilitation sessions. The conventional physiotherapy program will follow standard rehabilitation protocols and will include a structured stretching regimen comprising a 5-minute warm-up, 20 minutes of lower-limb stretching exercises, and a 5-minute cool-down.
  Interventions: Other: Vibration; Behavioral: Conventional Physical Therapy
- Group B (Near-Infrared Light + Conventional Physical Therapy) (Experimental): Participants allocated to this group will receive near-infrared (NIR) light therapy in addition to conventional physiotherapy. Near-infrared light will be applied to the lower limbs for 10 minutes during supervised rehabilitation sessions using a standardized therapeutic device. The conventional physiotherapy program will follow standard rehabilitation protocols and will include a structured stretching regimen consisting of a 5-minute warm-up, 20 minutes of lower-limb stretching exercises, and a 5-minute cool-down.
  Interventions: Other: Near-Infrared Light Therapy; Behavioral: Conventional Physical Therapy
- Group C ( (Infrared light + Vibration and Conventional Therapy) (Experimental): Participants allocated to this group will receive combined near-infrared (NIR) light therapy and vibration therapy in addition to conventional physiotherapy. Near-infrared light therapy will be applied to the lower limbs for 10 minutes using a standardized therapeutic device, followed by localized vibration therapy applied to the calf muscles for 10 minutes using a low-voltage vibration device during supervised rehabilitation sessions. The conventional physiotherapy program will follow standard rehabilitation protocols and will include a structured stretching regimen consisting of a 5-minute warm-up, 20 minutes of lower-limb stretching exercises, and a 5-minute cool-down.
  Interventions: Other: Near-Infrared Light Therapy; Other: Vibration; Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Other: Near-Infrared Light Therapy — The Near-infrared light therapy will be applied under the supervision of a qualified physiotherapist. Near-infrared light therapy involves the application of infrared lamps to the lower limbs to improve blood flow, reduce inflammation, and modulate neural activity associated with Restless Leg Syndrome symptoms. Participants in this group will receive NIR therapy for 10 minutes per session as part of the combined intervention. The intervention will be delivered three times per week for a total duration of 4 weeks.
  Arms: Group B (Near-Infrared Light + Conventional Physical Therapy); Group C ( (Infrared light + Vibration and Conventional Therapy)
Other: Vibration — Vibration therapy will be delivered using a low-voltage vibration device applied to the calf muscles. The therapy is intended to stimulate sensory receptors, improve neuromuscular function, and reduce symptom severity. Participants will receive vibration therapy for 10 minutes per session. The intervention will be delivered three times per week for a total duration of 4 weeks.
  Arms: Group A( Vibration Therapy + Conventional Physical Therapy); Group C ( (Infrared light + Vibration and Conventional Therapy)
Behavioral: Conventional Physical Therapy — The stretching program will be 30 minutes long, starting with a 5-minute warm-up, followed by 20 minutes of stretching exercises. The exercises will include hip rotation, quadriceps stretch, knee to chest stretch, hamstring stretch, gluteal stretch, straight leg raise, and side-lying leg lift. Each stretch will be held for 5 seconds and repeated for 3 sets of 10 repetitions.

SUMMARY:
This Randomized Clinical Trial, titled "Combined Effects of Near-Infrared Light and Vibration on Pain, Sleep Quality and Symptom Severity in Diabetic Patients with Restless Leg Syndrome," aims to evaluate a non-pharmacological treatment for Restless Leg Syndrome (RLS) in diabetic patients. RLS is a neurological disorder causing an irresistible urge to move the legs, and its co-occurrence with diabetes significantly worsens symptoms, pain, and sleep quality. While both Near-Infrared (NIR) light therapy and vibration therapy have individually shown benefits, this study will investigate the potential synergistic effects of combining them. 42 diabetic patients with RLS (aged 50-65) will be randomly assigned to one of three groups for four weeks (3 sessions/week): Group A (Vibration + Conventional Stretching), Group B (NIR Light + Conventional Stretching), and Group C (Combined Vibration and NIR Light + Conventional Stretching). Outcomes will be measured at baseline, 4 weeks, and 6 weeks using the International Restless Leg Syndrome Rating Scale (IRLS), the Pittsburgh Sleep Quality Index (PSQI), and the Numeric Pain Rating Scale (NPRS). This research explores the synergistic effects of near-infrared light and vibration therapy on Restless Leg Syndrome (RLS) symptoms in diabetic patients, aiming to alleviate symptoms, improve sleep quality, and enhance overall well-being.

DETAILED DESCRIPTION:
Restless Leg Syndrome (RLS) is a prevalent neurological sensorimotor disorder characterized by an uncontrollable urge to move the legs, often accompanied by uncomfortable sensations that worsen during rest and at night, leading to significant sleep disturbances and reduced quality of life. The condition is particularly common among individuals with diabetes, where peripheral neuropathy, poor glycemic control, and microvascular complications further exacerbate symptom severity. In Pakistan, evidence suggests a notably high prevalence of RLS in patients with type II diabetes, highlighting the clinical and public health importance of effective, context-specific management strategies. Although pharmacological treatments are commonly used, their side effects and limited long-term effectiveness emphasize the need for safe and sustainable non-pharmacological interventions.

Recent advances in physical therapy and rehabilitative care have increasingly focused on non-invasive sensory and neuromodulatory approaches to manage RLS symptoms. Near-infrared (NIR) light therapy and vibration therapy have independently demonstrated beneficial effects in reducing pain, improving peripheral circulation, decreasing symptom severity, and enhancing sleep quality in patients with RLS. However, existing studies are limited by small sample sizes, heterogeneous protocols, and a lack of long-term follow-up, particularly in diabetic populations. Importantly, despite encouraging individual results, the combined therapeutic effects of NIR light and vibration have not yet been systematically explored in diabetic patients with RLS, representing a significant gap in current rehabilitation research.

This randomized clinical trial aims to investigate the combined effects of near-infrared light and vibration therapy on pain intensity, sleep quality, and symptom severity in diabetic patients diagnosed with Restless Leg Syndrome. Participants meeting established diagnostic criteria will be recruited from multiple clinical settings and randomly allocated into three groups: vibration therapy with conventional stretching exercises, near-infrared light therapy with conventional stretching exercises, and a combined intervention group receiving both vibration and NIR therapy alongside conventional physiotherapy. Outcomes will be assessed at baseline, post-intervention, and follow-up using validated tools including the International Restless Legs Syndrome Rating Scale, Pittsburgh Sleep Quality Index, and Numeric Pain Rating Scale.

The findings of this study are expected to provide clinically meaningful evidence regarding the effectiveness of combined vibration and near-infrared light therapy as a non-pharmacological treatment approach for RLS in diabetic patients. By addressing pain, sleep disturbances, and symptom severity simultaneously, this combined intervention may offer a safer and more effective alternative to medication-dependent management. The results have the potential to inform clinical practice, support patient-centered rehabilitation strategies, and improve overall quality of life for individuals living with diabetes and Restless Leg Syndrome, particularly in resource-limited healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

Patients of age 50-65 years Both male and female patients with Type II diabetes Patients with a diagnosis of diabetes at least 6 months ago RLS (score of 11+ on the RLS scale) Patients meeting the four key RLS diagnosis criteria will be included in the study.

Criterion is: Urge to move due to uncomfortable leg sensations, symptoms worsening at rest, symptoms relief with movement ,greater symptom severity in the evening or at night.

Willingness to provide informed consent .

Exclusion Criteria:

Patients using analgesics, psychiatric, or neurological medications. Patients with any malignancies, neurological, skeletal, or vascular disorders History of drug abuse. Ongoing RLS treatments (e.g. vibration therapy, massage). Severe cognitive impairment. Pregnancy or lactation. Conditions contraindicating NIR or vibration therapy

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-14 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Rating Scale (IRLS) | Baseline, at 4th week, after 6th week
  Severity of Restless Leg Syndrome symptoms will be assessed using the International Restless Legs Syndrome Rating Scale (IRLS), a validated 10-item questionnaire designed to evaluate symptom severity and impact on daily life. Each item is scored on a 5-point Likert scale, with total scores ranging from 0 to 40, where higher scores indicate greater symptom severity. Improvement will be defined as a reduction in IRLS total scores following the intervention.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, at 4th week, after 6th week
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), a standardized 19-item self-report questionnaire assessing sleep quality and disturbances over the previous month. The global PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality. Improvement will be defined as a reduction in PSQI global scores following the intervention period.
Numeric Pain Rating Scale (NPRS) | Baseline, at 4th week, after 6th week
  Pain intensity associated with Restless Leg Syndrome will be evaluated using the Numeric Pain Rating Scale (NPRS). Participants will rate their pain on a scale from 0 (no pain) to 10 (worst imaginable pain). Improvement will be defined as a decrease in NPRS scores after completion of the intervention.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ratnani G, Harjpal P. Advancements in Restless Leg Syndrome Management: A Review of Physiotherapeutic Modalities and Their Efficacy. Cureus. 2023 Oct 10;15(10):e46779. doi: 10.7759/cureus.46779. eCollection 2023 Oct. PMID 37954781
- [Result] Ning P, Mu X, Yang X, Li T, Xu Y. Prevalence of restless legs syndrome in people with diabetes mellitus: A pooling analysis of observational studies. EClinicalMedicine. 2022 Mar 24;46:101357. doi: 10.1016/j.eclinm.2022.101357. eCollection 2022 Apr. PMID 35345532
- [Result] Coban O, Un Yildirim N, Yasa ME, Sonkaya AR. Effects of Different Exercise Programs on Symptoms, Sleep, and Quality of Life in Patients with Primary Restless Legs Syndrome. Mov Disord Clin Pract. 2023 Jul 27;10(9):1349-1359. doi: 10.1002/mdc3.13833. eCollection 2023 Sep. PMID 37772295